CLINICAL TRIAL: NCT00155883
Title: Bi-Weekly Docetaxel Plus 24-Hour Infusion of High-Dose 5-Fluorouracil / Leucovorin (HDFL) for Inoperable Advanced or Metastatic Gastric Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow a accrul due to many competitive trials.
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 921101
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2005-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: Taxteral
Drug: 5-Fluorouracil
Drug: Leucovorin

SUMMARY:
The primary objective is to determine the tumor response rate of bi-weekly docetaxel plus 24-hour infusion of high-dose 5-FU/leucovorin chemotherapy for patients with inoperable advanced gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer is one of the leading causes of cancer death in Taiwan. We have previously demonstrated that weekly 24-hour infusion of high-dose 5-fluorouracil (5-FU) and leucovorin is an effective and well-tolerated regimen for patients with advanced gastric cancer. Our in vitro and clinical studies suggested that long (24 hours or more) infusion of 5-FU/leucovorin may, compared with the conventional bolus regimens, enhance its anti-tumor activity in gastric cancer by prolonging suppression of thymidylate synthase, the target enzyme of 5-FU cytotoxicity. Docetaxel, a mitotic inhibitor, has good single-agent activity against gastric cancer, with a tumor response rate around 20 to 24%. Preliminary clinical data indicate that a biweekly administration of docetaxel will reduce the incidence of neutropenia and asthenia, two most bothersome side effects of tri-weekly and weekly docetaxel, respectively, while maintaining its anti-tumor activity. This phase II trial is designed to test the efficacy and toxicity of biweekly docetaxel and 24-hour infusion of high-dose 5-FU/leucovorin as first-line therapy for patients with inoperable advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven and inoperable advanced gastric adenocarcinoma.
2. Bi-dimensionally measurable disease by physical examination or image study (roentgenogram or computed tomography scan). The index lesions should be at least 20 mm × 10 mm in size.
3. Age must be older than 18 and younger than 75 year-old.
4. Karnofsky performance status>60% (see Appendix)
5. Adequate bone marrow reserves, defined as white blood cell (WBC)>4,000/l, absolute neutrophil count (ANC)>1,500/l, platelet>100,000/l.
6. Liver transaminases <2.5 times upper normal limit if no liver metastasis and 5 times upper normal limit if liver metastasis is present; total bilirubin <1.5 mg/dl; serum creatinine<1.5mg/dl.
7. Serum triglyceride level>70mg/dl.
8. Previous chemotherapy for metastatic disease is not allowed in this study. Previous adjuvant chemotherapy following curative gastrectomy is acceptable if the adjuvant chemotherapy has been completed for more than 6 months before enrollment into the present study.
9. Previous radiotherapy is allowed if the treatment was completed at least 4 weeks before the enrollment into this study.
10. Patients of childbearing age should have effective contraception during the study period.
11. All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional guidelines.

Exclusion Criteria:

1. Patients who are receiving concurrent radiotherapy, chemotherapy or other experimental therapy.
2. Patients who refuse port-A catheter implantation.
3. Patients with brain or leptomeningeal metastases.
4. Patients who have significant cardiac arrhythmia or acute myocardial infarction within 6 months before entry.
5. Patients who have major systemic diseases that the attending physicians considered inappropriate for systemic chemotherapy.
6. Life expectancy of less than 2 months.
7. Pregnant or nursing women may not participate. Women or men with reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
8. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancers, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any cancer from which the patient has been disease-free for 5 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2004-06; Study Completion 2005-07 (Estimated)

PRIMARY OUTCOMES:
tumor response rate

SECONDARY OUTCOMES:
clinical benefit response, toxicities, quality of life, time to disease progression, overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Lii Cheng, Study Chair — Department of Oncology , National Taiwan University Hospital; Ann-Lii Cheng, Principal Investigator — Department of Oncology, National Taiwan University Hospital
Locations (1):
- Department of Oncology, Nationa Taiwan University Hospital, Taipei, Taiwan